CLINICAL TRIAL: NCT06891846
Title: Evaluation of the Relationship Between Magnesium Depletion Score And Socket Healing Following Tooth Extraction
Brief Title: Relationship Between Magnesium Depletion Score and Extraction Socket Healing
Status: Completed | Type: Observational
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Sponsor
Other Study IDs: 24/738
Record Dates: First submitted 2025-02-04; First posted 2025-03-24 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-09

CONDITIONS: Wound Healing; Magnesium Level; Wisdom Tooth Removal
Keywords: blood magnesium level; oral surgery; wound healing

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants aged between 18-75 from both sexes: Systemically healthy participants, aged between 18-75 from both sexes

SUMMARY:
The surgical extraction of an impacted tooth is one of the most common procedures in oral surgery. Following extraction, the tissue undergoes repair and regeneration through a process known as socket healing (SH).

SH is a complex and highly regulated biological process. Several local, surgical, and systemic factors can influence SH. This study aimed to evaluate the impact of the magnesium depletion score (MDS) on the socket healing following tooth extraction.

DETAILED DESCRIPTION:
The surgical extraction of impacted teeth is one of the most commonly performed procedures in the field of oral surgery. According to the American Dental Association (ADA), surgical extraction involves "the removal of a tooth that has either erupted or not into the mouth, which includes the removal of a mucoperiosteal flap and the trimming of a portion of the tooth and/or bone." Complications related to post-extraction wound healing-such as pain, swelling, bleeding, and infection-can pose significant challenges for both patients and surgeons. Optimal healing depends not only on the tissue itself but also on various local, surgical, and systemic factors, including but not limited to the patient's stress levels, oral hygiene, age, sex, overall health status, and nutrition, many of which may be beyond intervention or control. Consequently, there is growing interest in treatments that can enhance wound healing. Recent studies indicate that magnesium consumption may have a beneficial effect on the healing process.

ELIGIBILITY:
Inclusion Criteria:

* Systemically healthy adult participants who were scheduled to undergo surgical extraction of lower impacted third molars.

Exclusion Criteria:

* Refusal to consent
* Presence of chronic diseases
* Use of medications that affect wound healing (steroids, bisphosphonate, or immunosuppressives)
* Prior radiotherapy in the head and neck area
* Pregnancy
* Inability to self-evaluate, and inability to communicate verbally or in writing.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Systemically healthy adult participants from both sexes, who were scheduled to undergo surgical extraction of lower impacted third molars, with a physical status classified as ASA I according to the American Society of Anesthesiologists (ASA).
Sampling Method: Probability Sample
Enrollment: 111 (Actual)
Dates: Start 2025-09-10 (Actual); Primary Completion 2025-10-22 (Actual); Study Completion 2025-10-22 (Actual)

PRIMARY OUTCOMES:
Magnesium depletion score (MDS) | 6 weeks
  The MDS is calculated by aggregating four factors:
  1. Diuretic use: Current use of diuretics is assigned 1 point.
  2. PPI use: Current use of proton pump inhibitors (PPIs) is assigned 1 point.
  3. Kidney function:
     * If the estimated glomerular filtration rate (eGFR) is between 60 and 90 mL/(min · 1.73 m²), 1 point is assigned.
     * If the eGFR is less than 60 mL/(min · 1.73 m²), 2 points are assigned.
  The total MDS score ranges from 0 to 4, based on the accumulation of points from these factors.
Assessment of Wound healing (WH) | 6 weeks
  Wound Healing (WH) will be assessed by using a scale called Inflammatory Proliferative Remodeling (IPR) Scale. According to the scale, each phase of WH is scored based on the parameters, including edema, bleeding and swelling.
  The total score of the IPR scale ranges from 0 to 16; 0-4 indicates poor healing; 5-10, acceptable healing; and 11-16, excellent healing.

SECONDARY OUTCOMES:
Post-operative pain | 3 days
  Post-operative pain will be assessed using the Visual Analog Scale (VAS). Patients will be asked to rate their pain on a scale from 0 to 10, where 0 indicates no pain and 10 represents the worst imaginable pain.

CONTACTS AND LOCATIONS:
Locations (1):
- Sağlık Bilimleri Üniversitesi Tacirler Eğitim Vakfı Sultanbeyli Ağız ve Diş Sağlığı Hastanesi, Istanbul, Sultanbeyli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Ye L, Zhang C, Duan Q, Shao Y, Zhou J. Association of Magnesium Depletion Score With Cardiovascular Disease and Its Association With Longitudinal Mortality in Patients With Cardiovascular Disease. J Am Heart Assoc. 2023 Sep 19;12(18):e030077. doi: 10.1161/JAHA.123.030077. Epub 2023 Sep 8. PMID 37681518
- [Result] Xu Y, Qin Y, Lu H, Liu L, Huang W, Huang A, Ye Y, Shen H, Guo Z, Chen W. The magnesium depletion score is associated with increased likelihood of kidney stone disease among female adults. J Trace Elem Med Biol. 2024 Jul;84:127432. doi: 10.1016/j.jtemb.2024.127432. Epub 2024 Mar 12. PMID 38489922
- [Result] Wang J, Xing F, Sheng N, Xiang Z. Associations of the Dietary Magnesium Intake and Magnesium Depletion Score With Osteoporosis Among American Adults: Data From the National Health and Nutrition Examination Survey. Front Nutr. 2022 May 31;9:883264. doi: 10.3389/fnut.2022.883264. eCollection 2022. PMID 35711538
- [Result] Fan L, Zhu X, Rosanoff A, Costello RB, Yu C, Ness R, Seidner DL, Murff HJ, Roumie CL, Shrubsole MJ, Dai Q. Magnesium Depletion Score (MDS) Predicts Risk of Systemic Inflammation and Cardiovascular Mortality among US Adults. J Nutr. 2021 Aug 7;151(8):2226-2235. doi: 10.1093/jn/nxab138. PMID 34038556
- [Result] Chen Y, Xiang X, Wu Y, Han S, Huang Z, Wu M. Magnesium Depletion Score Predicts Diabetic Retinopathy Risk among Diabetes: Findings from NHANES 2005-2018. Biol Trace Elem Res. 2023 Jun;201(6):2750-2756. doi: 10.1007/s12011-022-03384-3. Epub 2022 Aug 22. PMID 35989402